CLINICAL TRIAL: NCT02726841
Title: Superiority Trial of Type b Aortic Dissection Treatment Combined With Implantation of Bare Metal Stent in Abdominal Part of Aorta Versus Conventional Type b Treatment
Brief Title: Hybrid Treatment of Type B Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Dmitry Sirota, Cardiac surgeon, Meshalkin Research Institute of Pathology of Circulation
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAAD+bare stent
Record Dates: First submitted 2016-01-27; First posted 2016-04-04 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Aortic Dissection Type B
Keywords: Thoracic aorta; Abdominal aorta; Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid TAAD repair (Experimental): The group includes patients who underwent open thoracoabdominal aortic repair + abdominal stenting.
  Interventions: Procedure: Open thoracoabdominal aortic repair + abdominal stenting
- Conventional TAAD repair (Active Comparator): The group includes patients who underwent classic thoracoabdominal aortic repair with dacron prosthesis.
  Interventions: Procedure: Classic thoracoabdominal aortic repair

INTERVENTIONS:
Procedure: Open thoracoabdominal aortic repair + abdominal stenting — Thoracoabdominal aortic dissection (TAAD) repair + bare aortic stent (Djumbodis) implantation
  Other Names: Hybrid thoracoabdominal aortic repair
  Arms: Hybrid TAAD repair
Procedure: Classic thoracoabdominal aortic repair — Thoracoabdominal aortic dissection (TAAD) repair
  Other Names: Conventional TAAD repair
  Arms: Conventional TAAD repair

SUMMARY:
Authors hypothesize that thoracoabdominal aortic repair combined with bare metal stent implantation is superior over standard thoracoabdominal aortic repair.

DETAILED DESCRIPTION:
Main hypothesis of this study is that thoracoabdominal aortic repair combined with bare metal stent implantation is better permanent neurological deficits, perioperative bleeding, malperfusion of viscera over conventional thoracoabdominal aortic repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic aortic dissection type B
* Aortic size in descending thoracoabdominal aorta (TAA) > 55 mm

Exclusion Criteria:

* concomitant cardiac pathology
* concomitant oncology diseases in the last 5 years
* acute aortic dissection
* aortic size in visceral zone >45 mm
* connectivity tissue diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Permanent neurological events | 30 days
  Quantity of permanent neurological events such as stroke and paraplegia by 30th day after procedure.

SECONDARY OUTCOMES:
Perioperative bleeding | 5 days after procedure
  Volume of perioperative and postoperative bleeding in ICU
Mortality | 6 months
  Postoperative mortality will be measured during 6 months after procedure
Visceral malperfusion | 6 months
  Clinical evidences of visceral malperfusion (acute or achronic abdomen ischemia) during 6 months after procedure (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. Chernyavskiy, MD PhD, Study Chair — Academician Ye. Meshalkin Novosibirsk Research Institute of Circulation Pathology Ministry of Health care of Russian Federation

IPD SHARING:
Plan to Share IPD: No